CLINICAL TRIAL: NCT07012122
Title: Effect of Disturbed Attention on Balance in Children With Spastic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Abd Elnaser Abdelrahman, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/003969
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group of visual spatial memory task: It will consist of 21 children, who will perform a visual spatial memory task.
  Interventions: Other: visual spatial memory task
- Group of nonspatial verbal memory task: It will consist of 21 children, who will perform a nonspatial verbal memory task.
  Interventions: Other: nonspatial verbal memory task
- Group of visuomotor tracking task: It will consist of 21 children, who will perform a visuomotor tracking task.
  Interventions: Other: visuomotor tracking task

INTERVENTIONS:
Other: visual spatial memory task — The child will be asked to put numbers in an imagined matrices and memorize the position very well then will be asked to remember the position of these numbers.
  Groups: Group of visual spatial memory task
Other: nonspatial verbal memory task — The child is presented with a series of sentences that are similar in structure and content, with only slight variations in elements such as the verb, subject, or object. The child's task is to remember and accurately recall these sentences. For example: The dog is running in the park, The cat is running in the park, The dog is playing in the park, The dog is running in the yard.
  Groups: Group of nonspatial verbal memory task
Other: visuomotor tracking task — Then the rest will be introduced in the form of computer screen in front of the child with a dot moving under the control of a computer mouse and asking the child to track the dot while maintaining his balance as much as he can.
  Groups: Group of visuomotor tracking task

SUMMARY:
The purpose of the current study is to determine if there is a correlation between disturbed attention and balance in children with spastic diplegia.

DETAILED DESCRIPTION:
The neuromuscular impairments in children with cerebral palsy (CP) are manifested in abnormal posture and loss of selective motor control, poor trunk control and balance which contributes to poor postural control with significant limitations in their activities of daily living. Balance and upright postural control are fundamental components of movement which plays a major role in maintaining the body in equilibrium in a given sensory environment, with anticipatory and automatic postural adjustments. So, improving balance abilities in such children is fundamental.

In general, attention involves processes that allow individuals to focus on particular aspects of the environment and to mobilize sufficient effort for learning and problem solving.

Children with diplegic CP encounter difficulties in sensory processing and integration which influence the achievement of mature postural control.

There is reviews that didn't cover the relation between attention and balance. This study is to improve evidence regarding this area.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy children with spastic diplegia.
* Age ranges from 8 -12 years.
* Level Ι - II according to Gross Motor Functional Classification System (GMFCS).
* Grade 1, 1+ of the Modified Ashworth Scale.

Exclusion Criteria:

* Children that suffer from epilepsy.
* Severe visual and auditory problems.
* Structural or fixed soft tissue deformities of Lower extremities.
* Severe mental retardation.
* Botox injection in the lower extremity in the past 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sixty-three children with diplegic Cerebral Palsy of both genders that will be selected from Outpatient Clinic of Faculty of Physical Therapy, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Overall stability index (OSI) | One hour
  Values for the overall stability index (OSI) will be recorded by the Biodex balance system in the beginning with out any disturbance to the child attention, and then recorded during each task performed within their assigned group. Low OSI value indicates good balance and stability, with minimal sway or movement. High OSI value indicates difficulty maintaining balance and stability, with increased sway or movement, potentially suggesting impaired motor control or balance problems.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Osama Sayed, PhD, Study Chair — Assistant Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt